CLINICAL TRIAL: NCT02381353
Title: Postoperative Pain Control After Enucleation or Evisceration, a Double-Masked Randomized Controlled Trial of Standard Versus Slow-release Bupivacaine
Brief Title: Exparel Injection for Postoperative Orbital Pain
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth A. Bradley, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14-007145; NCT03003741 (obsolete NCT alias)
Record Dates: First submitted 2015-02-11; First posted 2015-03-06 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative
Keywords: Enucleation; Evisceration; Exparel; bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plain bupivacaine (Active Comparator): Intraoperative injection of local anesthetic agent, standard of care
  Interventions: Drug: Bupivacaine
- Exparel (sustained release bupivacaine) (Experimental): Intraoperative injection of local anesthetic agent, long acting agent
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Intraoperative orbital injection of local pain medication
  Other Names: Exparel

SUMMARY:
After surgery to remove the eye, either by enucleation or evisceration, patients have variable levels of pain for several postoperative days. Some patients have almost no discomfort while others require significant amounts of oral narcotics and report pain of 10 out of 10 on a numerical rating scale. The current operative standard is to infiltrate the eye socket with 0.5% bupivacaine during surgery leading to several hours of postoperative analgesia. In 2011, Pacira Pharmaceuticals released a bupivacaine liposomal injectable suspension (Exparel, 1.3%) which offers sustained release of bupivacaine giving postoperative pain control for up to 72 hours. This medication has been used in numerous surgeries including inguinal hernia repair, hemorrhoidectomy, bunionectomy, breast reconstruction, and orthopedic surgery, and the literature reports improved pain control, decreased use of oral opioids, and increased patient satisfaction. There are no reports of the use of Exparel in the ophthalmic literature. The investigators propose a randomized, controlled trial to compare the postoperative pain control offered by sustained release bupivacaine to that offered by standard plain bupivacaine after enucleation or evisceration.

ELIGIBILITY:
Inclusion criteria:

1. All patients undergoing enucleation or evisceration of the eye whose surgery is performed by the Department of Ophthalmology at Mayo Clinic Rochester
2. Willing and able to comprehend a numerical rating scale system and provide a score to assess pain, nausea, and satisfaction level.

Exclusion criteria:

1. Age less than 18 years (Exparel has not been tested in a pediatric population)
2. Pregnant or nursing (Exparel has not been tested in this patient population)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative orbital pain | Days 3 postoperatively
  Pain on a scale of 0-10, assessed on day 3 post enucleation or evisceration

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | Days 3 postoperatively
  Nausea and vomiting on a scale of 0-3, assessed on day 3 post enucleation or evisceration
Quantity of oral narcotics used for postoperative pain control | Days 3 postoperatively
  Number of oral narcotic pills taken during postoperative days 0-3
Patient satisfaction | Day 3 postoperatively
  Overall satisfaction with postoperative recovery, assessed on a scale of 1-5
Postoperative complications | 6-8 weeks postoperatively
  Assessment of any postsurgical complications completed at postoperative visit

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bradley, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Michigan Kellogg Eye Institute, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
University of Michigan will share patient study data with Mayo site. A Data Use Agreement has been approved for this purpose.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From July 2024 through end of reporting period.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials